CLINICAL TRIAL: NCT06764498
Title: Retrospective Study to Evaluate the Effectiveness of the Approach to Enuresis in Our Center
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ENU-PED-21-02
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Enuresis
Keywords: Enuresis; Children
MeSH Terms: conditions — Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study to evaluate the effectiveness of the approach to enuresis at IRCCS Azienda Ospedaliero-Universitaria of Bologna Policlinico di Sant'Orsola, Italy.

DETAILED DESCRIPTION:
Enuresis is an extremely common condition that affects 5-10% of 7-year-olds and 3% of adolescents and persists in 2% of adults. Although in most cases it is not related to comorbidities and more serious illnesses, enuresis can have long-term negative impacts on the psychological sphere of both the children by leading to low self-esteem, anxiety, and embarrassment and the entire family by leading to stress and intolerance toward the condition and an overall reduction in quality of life.

Enuresis is defined as the involuntary loss of urine during sleep that occurs at least twice a week in a sleeping child older than 5 years. It is classified into primary, if the child has never achieved continence, or secondary if it appears after an enuresis-free period of at least 6 months. It can be further subdivided into monosymptomatic and non-monosymptomatic enuresis, the latter defined by the coexistence of daytime incontinence or lower urinary tract symptoms such as daytime incontinence, urgency, difficulty urinating, and low/high daytime urinary frequency.

There are multiple guidelines in the literature regarding the approach to be taken for the management of enuresis. In 2015 from a consensus among the leading international pediatric urology and nephrology societies, practical guidelines to the approach to the pediatric enuretic patient were developed.

Two main types of approach are proposed in this paper, one of which has been adopted in our center and represents a more scrupulous modality in that during the first visit, not only useful advice on good urination practices is given, but also two diaries, one "daily" which assesses the volume of fluid ingested, the amount of urine produced daily, and urinary leakage the other "nocturnal" through which parameters such as bladder capacity and the amount of urine produced during the night are investigated, which allow not only to distinguish between monosymptomatic and non-monosymptomatic enuresis, but also to provide an objective method on which to base the choice of possible therapy - alert or desmopressin - which is therefore not provided before a second clinical checkup. Given the large number of pediatric patients referred to our Center for the problem of enuresis, this study aims to analyze the effectiveness of the methodology adopted on the resolution of this condition.

The primary aim of this study is to assess the resolution rate of enuresis in our population. The secondary aims of this study are to evaluate the effectiveness of the proposed pharmacological treatments, and to evaluate the correlation between constipation and enuresis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex under the age of 18 years at the time of the first outpatient visit;
* Patients clinically evaluated in the outpatient clinic during the period 01/05/2019- 31/05/2021 with a diagnosis of enuresis;
* Patients presenting at least two outpatient follow-ups;
* Informed consent signed by parent or legal guardian.

Exclusion Criteria:

* Patients older than 18 years of age;
* Patients who lack completed night and daily diaries;
* Patients with continuous incontinence;
* Patients with neurological disorders and/or signs of spinal occult dysraphism;
* Patients with a severe cognitive disorder.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Since this is a descriptive study, a formal calculation of sample size is not expected. However, about 150-200 subjects are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily urinary frequency | at baseline
  increase (≥8 micturitions/day) or decrease (≤3 micturitions/day)
Maximum Voided Volume (MVV) | at baseline
  volume of urine emitted in 24 hours, excluding first morning urine
Bladder capacity | at baseline
  reduction (<35% of expected bladder capacity) or increase (> 150% of expected bladder capacity)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pasini, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy